CLINICAL TRIAL: NCT07249515
Title: ınvestigation of the Relationship Between Scapular Position and Upper Extremity Performance in Adolescents With Idiopathic Scoliosis
Brief Title: Scapula and Upper Extremity Performance in Scoliosis
Status: Recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Tuğçe Yavuz, Principal Investigator, Istinye University
Other Study IDs: 25-120
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Adolescent Idiopathic Scoliosis; Upper Extremity
Keywords: Adolescent Idiopathic Scoliosis; Performance; Scapula; upper extremity performance
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescent Idiopathic Scoliosis Group: Participants with Adolescent Idiopathic Scoliosis underwent assessments of scapular dyskinesis, scapular lateral displacement, and upper extremity performance using standardized functional tests.
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Participants with Adolescent Idiopathic Scoliosis underwent assessments of scapular dyskinesis, scapular lateral displacement, and upper extremity performance using standardized functional tests.

SUMMARY:
Adolescent Idiopathic Scoliosis s a three-dimensional spinal deformity that may alter shoulder girdle alignment, scapular orientation, and upper extremity biomechanics. Changes in scapular position can influence arm movement, muscle activation, and overall functional performance. Understanding these relationships is clinically important for developing effective exercise and rehabilitation strategies.

The aim of this study is to examine the association between scapular position and upper extremity performance in adolescents diagnosed with Adolescent Idiopathic Scoliosis. Scapular dyskinesis, scapular lateral displacement, and upper limb functional performance will be evaluated and correlated with Cobb angle severity. Findings may help clinicians better understand functional impairments linked to scoliosis and support more targeted rehabilitation programs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Adolescent Idiopathic Scoliosis
* Age 10-19 years
* Cobb angle between 10° and 45°
* No prior scoliosis-specific conservative treatment
* Ability to participate in physical assessments
* Voluntary willingness to participate

Exclusion Criteria:

* Neuromuscular, congenital, or syndromic scoliosis
* Prior spinal surgery
* Shoulder injury or upper limb pathology affecting performance
* Neurological or rheumatological disorders
* Communication or cognitive limitations interfering with testing

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of adolescents aged 10 to 19 years who have been clinically and radiographically diagnosed with Adolescent Idiopathic Scoliosis. Participants must have a Cobb angle between 10° and 45°, no previous scoliosis-specific conservative treatment, and the physical ability to complete scapular assessment and upper extremity performance testing.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Medicine Ball Throw Test | 4 weeks
  The test will be used to assess upper extremity explosive power. Participants will be positioned in an upright chair without armrests, with their ankles, knees, and hips at 90 degrees. They will be asked to grasp a 3-kg medicine ball with both hands and throw it overhead without bending their bodies forward or flexing their elbows. The first point where the ball touches the floor will be measured from the starting point, and the value will be recorded in cm. The test will be repeated three times, and the average will be recorded. If participants throw the ball down to neck level or by bending forward from the body, the test will be invalid and the test will be repeated.

SECONDARY OUTCOMES:
Scapular Dyskinesis Test | 4 weeks
  This is a dynamic test in which the individual, using weights determined by the individual's body weight, actively abducts and flexes their arms bilaterally and with the weight in hand. These movements are repeated several times, and scapular winging, scapular asymmetry, and abnormal movements during these movements indicate the presence of scapular dyskinesis. The type of scapular dyskinesis is determined after these repetitions.
Scapular Lateral Slip Test | 4 weeks
  The Scapular Lateral Slip Test, as defined by Kibler, is a semi-dynamic test commonly used to assess the presence of scapular dyskinesis. The individual to be tested was assessed in a standing position with their back turned and open. In the test performed to assess dominant and non-dominant scapular positions, the distance between the spinous process of the T3 vertebra and the medial end of the scapula root (spinal root) and the distance between the spinous process of the T7 vertebra and the inferior end of the scapula were measured with a tape measure and recorded in centimeters (cm). A difference of more than 1.5 cm between the dominant and non-dominant side measurements indicates a positive test.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No